CLINICAL TRIAL: NCT02769299
Title: Cardiotoxicity of Radiation Therapy (CTRT)
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 04115
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer; Lung Cancer; Mediastinal Lymphomas
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: Radiation Therapy — less than 1 Gy with protons to 4-8 Gy with photons

SUMMARY:
The overall objective of this proposal is to determine the utility of sensitive imaging and biomarker measures in detecting subclinical cardiotoxicity across a spectrum of radiation doses to the heart. We will focus specifically on patients receiving photon or proton chest radiotherapy. Our broad working hypothesis is that RT induces early, subclinical CV injury, as evidenced by cardiomyocyte inflammation and necrosis, and worsening CV function.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Patients with left sided breast cancer newly initiating fractionated whole breast/chest wall with regional nodal photon or proton radiation therapy.
* Patients with right sided breast cancer with newly initiating fractionated photon or proton radiation therapy with mediastinal nodal proton or photon radiation therapy that will include cardiac dose.
* Lung cancer patients treated with definitive intent (greater than or equal to 50 Gy) using fractionated thoracic radiotherapy with proton or photon radiation therapy. Patients receiving concurrent chemotherapy will be allowed.
* Patients with mediastinal lymphoma, whose lowest extent of mediastinal disease is at or below the level of the carina, treated with consolidative radiation with definitive intent (greater than or equal to 20 Gy) using fractionated thoracic radiotherapy with proton or photon radiation therapy.
* Ability to read and comprehend English.

Exclusion Criteria:

* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Patients receiving stereotactic body radiotherapy
* Patients unable to undergo MR imaging will be excluded from the optional MR, but will not be excluded from the main study.
* Life expectancy less than 12 months
* Vulnerable patients as noted in 5 below (children, pregnant women, fetuses, neonates, or prisoners)
* Patients with estimated glomerular filtration rate of less than 60 ml/min/1.73sq.m will be excluded from the optional MR, but will not be excluded from the main study.
* Non-diagnostic echocardiography windows

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: breast cancer, lung cancer, and mediastinal lymphomas
Sampling Method: Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2015-06-02 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
Number of CV injury | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Ky, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States